CLINICAL TRIAL: NCT00903617
Title: A Two Part, Multicenter Phase IIa, Placebo Controlled Study, to Examine the Safety, Tolerability, and Effects of GSK256073 on Lipids in Subjects With Dyslipidemia
Brief Title: Study to Test GSK256073 in Patients With Dyslipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112795
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Dyslipidaemias; Dyslipidemias
Keywords: lipids; HM74A
MeSH Terms: conditions — Dyslipidemias | interventions — 8-chloro-3-pentyl-1H-purine-2,6(3H,7H)-dione; Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A Treatment A (Experimental): 5 mg of GSK256073
  Interventions: Drug: GSK256073
- Part A Treatment B (Experimental): 50 mg of GSK256073
  Interventions: Drug: GSK256073
- Part A Treatment C (Experimental): 150 mg of GSK256073
  Interventions: Drug: GSK256073
- Part A Treatment D (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Part B Treatment A (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Part B Treatment B (Active Comparator): 1500 mg Niaspan
  Interventions: Drug: Niaspan
- Part B Treatment C (Experimental): x mg dose of GSK256073 based on data from Part A
  Interventions: Drug: GSK256073
- Part B Treatment D (Experimental): optional dose of GSK256073 based on data from Part A
  Interventions: Drug: GSK256073

INTERVENTIONS:
Drug: GSK256073 — 5 mg for 8 weeks
  Arms: Part A Treatment A
Drug: GSK256073 — 50 mg for 8 weeks
  Arms: Part A Treatment B
Drug: GSK256073 — 150 mg for 8 weeks
  Arms: Part A Treatment C
Drug: Placebo — placebo for 8 weeks
  Arms: Part A Treatment D; Part B Treatment A
Drug: Niaspan — 1500 mg for 8 weeks
  Arms: Part B Treatment B
Drug: GSK256073 — x mg for 8 weeks based from data from Part A
  Arms: Part B Treatment C
Drug: GSK256073 — optional dose based on data from Part A
  Arms: Part B Treatment D

SUMMARY:
This is a two part study (Part A and Part B) that will first aim to establish the PK/PD relationship between exposure and lipid effects (Part A: 75 subjects), and will then confirm the effect using the most relevant dose(s) (Part B: ~90 subjects). Doses of 5mg, 50mg and 150mg of GSK256073 will be administered in Part A, and the dose(s) for Part B will be based on the PK/PD data from Part A. Data from Part A and Part B will be combined to decrease overall subject numbers needed in part B. Part B of the study will include a niaspan arm for relative comparison of the effects of GSK256073 and niacin on lipids and flushing

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to beginning study-related procedures. Subjects must understand the aims, investigational procedures and possible consequences of the study and must be able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Male or female 18-75 years of age at screening.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea.
* Male subjects must agree to use one of several pre-specified contraception methods. This criterion must be followed from the time of the first dose of study medication until three days following the last dose.
* Body weight > 50 kg (110 pounds) and body mass index (BMI) between 19 and 39 (inclusive)
* LDLc concentration ≥100 mg/dL at screening and within 4 weeks of randomization (if screening occurs > 4 weeks prior to randomization)
* Fasting triglyceride concentration ≤ 300 mg/dL at screening and within 4 weeks of randomization (if screening occurs > 4 weeks prior to randomization)
* HDLc ≤ 45 mg/dL for males or ≤ 55 mg/dL for females at screening and within 4 weeks of randomization (if screening occurs > 4 weeks prior to randomization)
* Subject currently receiving lipid-modifying medication(s) must agree to stop medication(s) for at least 6 weeks prior to randomization. After this washout period LDL, TG and HDL values must be remeasured and meet the above criteria prior to randomization in the study
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Evidence of clinical instability based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk and will not interfere with the study procedures.
* Any change in concomitant medication (including multivitamins, herbal remedies, dietary supplements, and over-the-counter medication) within six weeks prior to screening that is not approved by GSK.
* Any change in diet, exercise habits or smoking status within six weeks prior to screening.
* A medical history significant for the following:
* Clinical cardiovascular disease, including history or current evidence of coronary heart disease, heart failure, cerebrovascular disease, peripheral vascular disease, and/or a 10-year risk of CHD > 20% while on or titrated off lipid lowering medication. Subjects pending diagnostic procedures for any of those conditions at the time of screening will not be eligible for participation.
* Renal impairment (for males) as defined by a calculated GFR < 60 mL/min . Renal impairment (for females) as defined by a calculated GFR < 55 ml/min.
* History of diabetes mellitus, or history of post-prandial and/or random blood glucose > 200 mg/dl or fasting glucose > 125 mg/dL or currently taking diabetes medications to manage fasting glucose levels (e.g. glitazones, sulfonylureas, insulin, metformin, etc.).
* History of anemia or treatment of anemia within 12 months of screening or Hgb or Hct below the lower limit of reference range for age and gender at screening
* History of pancreatitis
* Any concurrent serious illness (e.g., severe COPD, HIV positive, liver cirrhosis, history of malignancy other than skin cancer within 5 years of initial diagnosis or with evidence of recurrence) that may interfere with a subject from completing the study
* Active peptic ulcer disease (PUD) and/or history of PUD or other gastrointestinal bleeding within 12 months prior to screening.
* History of kidney stones
* History of gout and/or hyperuricemia or taking drugs for hyperuricemia: allopurinol and/or probenecid
* History of Gilbert's syndrome
* Current inadequately controlled hypertension (blood pressure ≥160 mmHg systolic or ≥100 mmHg diastolic at screening). If blood pressure medication is changed, blood pressure will be re-measured after 6 weeks and must again meet these criteria.
* An unwillingness of subjects currently taking aspirin to reduce the daily dose to 81 mg starting 2 weeks prior to first dose and until the follow-up visit.
* Creatinine phosphokinase (CPK) 2X ULN at screening.
* A serum uric acid exceeding by ≥ 15% the upper limit of the reference range at screening.
* PT and/or aPTT above the reference range.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has a positive pre-study drug screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Use of the following blood pressure medications is prohibited at any dose: enalapril, losartan, captopril
* If subjects are titrated or switched to alternative therapy they must be on a stable dose for at least 4 weeks prior to randomization.
* Subjects will be excluded if they require treatment with systemic corticosteroids
* Subjects will be excluded if they take quinolone antibiotics, methotrexate, ibuprofen or other medication secreted by renal OAT transporters
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to dosing
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* History of sensitivity or untoward reaction to the study medications (i.e. GSK256073 or Niaspan), or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.
* A positive test for HIV antibody.
* Subject is mentally or legally incapacitated.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-06-15 (Actual); Primary Completion 2010-02-16 (Actual); Study Completion 2010-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (11):
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Brooklyn Center, Minnesota
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Olympia, Washington
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20061

REFERENCES:
- [Background] Olson EJ, Mahar KM, Haws TF, Fossler MJ, Gao F, de Gouville AC, Sprecher DL, Lepore JJ. A Randomized, Placebo-Controlled Trial to Assess the Effects of 8 Weeks of Administration of GSK256073, a Selective GPR109A Agonist, on High-Density Lipoprotein Cholesterol in Subjects With Dyslipidemia. Clin Pharmacol Drug Dev. 2019 Oct;8(7):871-883. doi: 10.1002/cpdd.704. Epub 2019 Jul 3. PMID 31268250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 centers in the United States from 15 June 2009 to 16 February 2010.
Pre-assignment Details: A total of 80 participant were enrolled in the study. Participants on lipid-altering medications (prescription, over-the-counter and herbal preparations directed at lipid lowering) were washed out of their treatment for at least 6 weeks prior to randomization and 8 weeks wash out for participants on fibrate medications.
Groups:
- GSK256073 5 mg: Eligible participants received GSK256073 5 milligrams (mg) oral tablet once daily for 60 days. Participants were provided study medication at the Baseline/randomization Visit. Study medication was self administered each morning (in a fed state) for 60 consecutive days during the out-patient visit. Participant were given a new supply of study medication approximately every 2 weeks at the out-patient visits.
- GSK256073 50 mg: Eligible participants received GSK256073 50 mg oral tablet once daily for 60 days. Participants were provided study medication at the Baseline/randomization Visit. Study medication was self administered each morning (in a fed state) for 60 consecutive days during the out-patient visit. Participant were given a new supply of study medication approximately every 2 weeks at the out-patient visits.
- GSK256073 150 mg: Eligible participants received GSK256073 150 mg oral tablet once daily for 60 days. Participants were provided study medication at the Baseline/randomization Visit. Study medication was self administered each morning (in a fed state) for 60 consecutive days during the out-patient visit. Participant were given a new supply of study medication approximately every 2 weeks at the out-patient visits.
- Placebo: Eligible participants received placebo matching GSK256073 oral tablet once daily for 60 days. Participants were provided study medication at the Baseline/randomization Visit. Study medication was self administered each morning (in a fed state) for 60 consecutive days during the out-patient visit. Participant were given a new supply of study medication approximately every 2 weeks at the out-patient visits.
Period: Overall Study
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Started | 19 | 20 | 20 | 21
Completed | 16 | 15 | 15 | 20
Not Completed | 3 | 5 | 5 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Protocol-defined stopping criteria | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK256073 5 mg: Eligible participants received GSK256073 5 mg oral tablet once daily for 60 days. Participants were provided study medication at the Baseline/randomization Visit. Study medication was self administered each morning (in a fed state) for 60 consecutive days during the out-patient visit. Participant were given a new supply of study medication approximately every 2 weeks at the out-patient visits.
- Total: Total of all reporting groups
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo | Total
Number analyzed (Participants) | 19 | 20 | 20 | 21 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (8.43) | 53.8 (9.77) | 57.0 (10.75) | 57.7 (10.15) | 56.7 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 11 | 41
  Male | 9 | 10 | 10 | 10 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 18 | 18 | 19 | 18 | 73
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The GSK256073 Area Under Concentration-time Curve (AUC) and High Density Lipoprotein Cholesterol (HDLc) Data to Evolve the Exposure-response Pharmacokinetic/Pharmacodynamic (PK/PD) Relationship for Changes in HDLc Levels
Description: The potential PK/PD relationship was to be assessed by plotting GSK256073 AUCs against HDLc. The PK/PD model that was to be used for the simulations in the study design was to be refined with the Part A observed AUC exposures and HDLc levels. However, the study was stopped for futility at the end of Part A due to lack of a compelling PK/PD relationship between GSK256073 and lipid effects that would predict success in achieving significant HDLc raising.
Time Frame: Week 2, 4, 6 and 8
Population: Data was not collected as the study was stopped for futility at the end of Part A due to lack of a compelling PK/PD relationship between GSK256073 and lipid effects that would predict success in achieving significant HDLc raising.
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect, medically significant or it is associated with liver injury and impaired liver function.
Time Frame: Up to follow up (14 days from last dose)
Population: Safety Population was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- GSK256073 50 mg: Eligible participants received GSK256073 5 mg oral tablet once daily for 60 days. Participants were provided study medication at the Baseline/randomization Visit. Study medication was self administered each morning (in a fed state) for 60 consecutive days during the out-patient visit. Participant were given a new supply of study medication approximately every 2 weeks at the out-patient visits.
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants
  Any AEs | 8 | 12 | 17 | 14
  Any SAEs | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Electrocardiography (ECG) Findings
Description: Single 12-lead ECGs was obtained at each time point during the study using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QTc intervals. Participants with normal, abnormal- clinically significant (CS) and abnormal- not clinically significant (NCS) ECG values were reported.
Time Frame: Up to Week 8
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants
  Baseline, Predose, Normal | 9 | 5 | 8 | 13
  Baseline, Predose, Abnormal-NCS | 10 | 15 | 12 | 8
  Baseline, Predose, Abnormal-CS | 0 | 0 | 0 | 0
  Week 2, Predose, Normal: number analyzed (Participants) | 18 | 19 | 19 | 20
  Week 2, Predose, Normal | 10 | 10 | 9 | 13
  Week 2, Predose, Abnormal-NCS: number analyzed (Participants) | 18 | 19 | 19 | 20
  Week 2, Predose, Abnormal-NCS | 8 | 9 | 10 | 7
  Week 2, Predose, Abnormal-CS: number analyzed (Participants) | 18 | 19 | 19 | 20
  Week 2, Predose, Abnormal-CS | 0 | 0 | 0 | 0
  Week 4, Predose, Normal: number analyzed (Participants) | 17 | 17 | 18 | 20
  Week 4, Predose, Normal | 8 | 5 | 10 | 16
  Week 4, Predose, Abnormal-NCS: number analyzed (Participants) | 17 | 17 | 18 | 20
  Week 4, Predose, Abnormal-NCS | 9 | 12 | 8 | 4
  Week 4, Predose, Abnormal-CS: number analyzed (Participants) | 17 | 17 | 18 | 20
  Week 4, Predose, Abnormal-CS | 0 | 0 | 0 | 0
  Week 6, Predose, Normal: number analyzed (Participants) | 16 | 16 | 16 | 20
  Week 6, Predose, Normal | 9 | 4 | 10 | 15
  Week 6, Predose, Abnormal-CS: number analyzed (Participants) | 16 | 16 | 16 | 20
  Week 6, Predose, Abnormal-CS | 7 | 12 | 6 | 5
  Week 6, Predose, Abnormal-NCS: number analyzed (Participants) | 16 | 16 | 16 | 20
  Week 6, Predose, Abnormal-NCS | 0 | 0 | 0 | 0
  Week 8, 0 hour, Normal: number analyzed (Participants) | 16 | 15 | 15 | 20
  Week 8, 0 hour, Normal | 10 | 5 | 9 | 13
  Week 8, 0 hour, Abnormal-NCS: number analyzed (Participants) | 16 | 15 | 15 | 20
  Week 8, 0 hour, Abnormal-NCS | 6 | 10 | 6 | 7
  Week 8, 0 hour, Abnormal-CS: number analyzed (Participants) | 16 | 15 | 15 | 20
  Week 8, 0 hour, Abnormal-CS | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Vital Signs-Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP was assessed at Baseline (Week 0), Week 2, 4, 6 and 8. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the post-Baseline value from the Baseline value.
Time Frame: Baseline (Week 0) up to Week 8
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Millimeters of mercury (mmHg)
  DBP, Week 2, 0 hour: number analyzed (Participants) | 18 | 19 | 19 | 20
  DBP, Week 2, 0 hour | -2.1 (6.39) | -0.1 (4.93) | -1.0 (3.42) | 1.1 (4.86)
  DBP, Week 4, 0 hour: number analyzed (Participants) | 17 | 17 | 18 | 20
  DBP, Week 4, 0 hour | -2.6 (3.97) | 0.8 (7.12) | 0.8 (3.61) | 1.6 (5.35)
  DBP, Week 6, 0 hour: number analyzed (Participants) | 16 | 16 | 16 | 20
  DBP, Week 6, 0 hour | -0.6 (5.37) | -1.3 (7.53) | 1.6 (5.51) | 1.4 (5.28)
  DBP, Week 8, 0 hour: number analyzed (Participants) | 16 | 15 | 15 | 20
  DBP, Week 8, 0 hour | 0.8 (6.41) | -1.7 (8.47) | 2.0 (6.89) | 1.9 (5.43)
  SBP, Week 2, 0 hour: number analyzed (Participants) | 18 | 19 | 19 | 20
  SBP, Week 2, 0 hour | -3.0 (11.03) | 2.7 (9.91) | -2.7 (5.54) | 2.1 (9.25)
  SBP, Week 4, 0 hour: number analyzed (Participants) | 17 | 17 | 18 | 20
  SBP, Week 4, 0 hour | -4.5 (11.27) | 6.1 (11.74) | -3.2 (5.17) | 4.2 (9.46)
  SBP, Week 6, 0 hour: number analyzed (Participants) | 16 | 16 | 16 | 20
  SBP, Week 6, 0 hour | 3.7 (9.86) | 0.9 (12.12) | -0.1 (10.21) | 0.2 (9.29)
  SBP, Week 8, 0 hour: number analyzed (Participants) | 16 | 15 | 15 | 20
  SBP, Week 8, 0 hour | 1.8 (10.64) | 1.0 (13.96) | -1.3 (8.35) | 0.8 (9.00)

5. Secondary Outcome: Change From Baseline in Vital Signs-Heart Rate
Description: Heart rate was assessed at Baseline (Week 0), Week 2, 4, 6 and 8. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the post-Baseline value from the Baseline value.
Time Frame: Baseline (Week 0) up to Week 8
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Beats per minute
  Week 2, 0 hour: number analyzed (Participants) | 18 | 19 | 19 | 20
  Week 2, 0 hour | 1.4 (8.14) | -0.5 (7.17) | 1.9 (4.21) | 1.1 (4.20)
  Week 4, 0 hour: number analyzed (Participants) | 17 | 17 | 18 | 20
  Week 4, 0 hour | -1.2 (4.82) | -1.9 (5.61) | 3.6 (4.83) | 1.9 (5.31)
  Week 6, 0 hour: number analyzed (Participants) | 16 | 16 | 16 | 20
  Week 6, 0 hour | -1.4 (6.85) | -0.2 (5.96) | 2.8 (4.97) | 3.6 (5.61)
  Week 8, 0 hour: number analyzed (Participants) | 16 | 15 | 15 | 20
  Week 8, 0 hour | 0.0 (7.25) | 3.5 (4.37) | 4.6 (5.87) | 2.2 (4.53)

6. Secondary Outcome: Number of Participants With Abnormal Hematology Values
Description: Blood samples for assessment of hematology parameters of platelet count, red blood cell count, white blood cell count, hemoglobin, haptoglobin, reticulocyte count, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, neutrophils, lymphocytes, monocytes, eosinophils and basophils was collected at Baseline and at Weeks 2, 4, 6 and 8.
Time Frame: Baseline (Week 0) up to Week 8
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Values
Description: Blood samples for assessment of clinical chemistry parameters of blood urea nitrogen, creatinine, glucose (fasting), sodium, creatine phosphokinase, potassium, chloride, total carbon dioxide, calcium, total lactose dehydrogenase (LDH), aspartate aminotransferase (AST), alanine amino transferase (ALT), gamma glutamyl transferase (GGT), alkaline phosphatase, phosphate, total and direct bilirubin, uric acid, albumin and total protein was collected at Baseline and at Weeks 2, 4, 6 and 8.
Time Frame: Up to Week 8
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants
  Creatine kinase, Week 6, High: number analyzed (Participants) | 16 | 16 | 16 | 20
  Creatine kinase, Week 6, High | 0 | 1 | 0 | 0
  Phosphorous, inorganic, Week 8, low: number analyzed (Participants) | 16 | 15 | 15 | 20
  Phosphorous, inorganic, Week 8, low | 1 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormal Urinalysis Results
Description: Urinalysis assessment was done for urine occult blood, urine glucose, urine ketones and urine protein over eight weeks treatment period.
Time Frame: Up to Week 8
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants
  Urine Occult Blood, Baseline, Predose, 1+ | 0 | 0 | 1 | 0
  Urine Occult Blood, Baseline, Predose, Trace | 0 | 1 | 0 | 1
  Urine Occult Blood, Week 2, Predose, 1+ | 0 | 0 | 1 | 0
  Urine Occult Blood, Week 2, Predose, Trace | 0 | 2 | 0 | 2
  Urine Occult Blood, Week 4, Predose, 1+ | 0 | 0 | 0 | 1
  Urine Occult Blood, Week 4, Predose, Trace | 0 | 1 | 1 | 0
  Urine Occult Blood, Week 6, Predose, 3+ | 0 | 0 | 1 | 0
  Urine Occult Blood, Week 6, Predose, Trace | 0 | 2 | 0 | 0
  Urine Occult Blood, Week 8, 0 hour, 1+ | 0 | 0 | 0 | 1
  Urine Occult Blood, Week 8, 0 hour, Trace | 0 | 0 | 2 | 0
  Urine Ketones, Baseline, Predose, Trace | 0 | 1 | 0 | 0
  Urine Ketones, Week 2, Predose, Trace | 0 | 0 | 1 | 0
  Urine Ketones, Week 4, Predose, 2+ | 0 | 0 | 1 | 0
  Urine Ketones, Week 6, Predose, Trace | 0 | 1 | 0 | 0
  Urine Ketones, Week 8, 0 hour, 1+ | 0 | 0 | 1 | 0
  Urine Protein, Baseline, Predose, Trace | 0 | 1 | 1 | 2
  Urine Protein, Week 2, Predose, Trace | 1 | 1 | 0 | 1
  Urine Protein, Week 4, Predose, 1+ | 0 | 0 | 1 | 0
  Urine Protein, Week 4, Predose, Trace | 0 | 1 | 2 | 0
  Urine Protein, Week 6, Predose, 1+ | 0 | 0 | 1 | 0
  Urine Protein, Week 6, Predose, Trace | 1 | 1 | 1 | 1
  Urine Protein, Week 8, 0 hour, 1+ | 0 | 0 | 0 | 1
  Urine Protein, Week 8, 0 hour, Trace | 1 | 0 | 3 | 2

9. Secondary Outcome: Average Global Flushing Score
Description: Flushing assessment was captured by participants in individual diaries provided to each study participant. Participants were instructed to return their diaries after each study visit (Week 2, Week 4, Week 6 and Week 8) where they were given a new diary for the time between visits. Flushing symptom questionnaire (FSQ) was used to measure participant reported feelings of severity associated with different types of flushing symptoms. The FSQ comprised of 11 items. The response scale combined verbal descriptors as well as a 0-10 numerical rating scale. Items 1, 2, 4 and 10 had verbal descriptors. The items 3, 5, 6, 7, 8, 9 and 11 were rated on a 0 to 10 scale (none=0, mild=1-3, moderate=4-6, severe=7-9 and extreme=10). The total score for these items ranged from 0 (not at all) to 70 (extreme). Higher score indicated more severe flushing symptoms and 0 indicated no flushing symptoms.
Time Frame: Up to Week 8
Population: PD Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants
  None | 15 | 16 | 8 | 15
  Mild | 2 | 2 | 8 | 4
  Moderate | 1 | 2 | 4 | 0
  Severe | 0 | 0 | 0 | 1

10. Secondary Outcome: Number of Participants With Self Reported Assessment of Flushing
Description: Flushing assessment was captured by participants in individual diaries provided to each study participant. Participants were instructed to return their diaries after each study visit (Week 2, Week 4, Week 6 and Week 8) where they were given a new diary for the time between visits. Participants were asked to perform an assessment of their perceived flushing intensity after their completion of VAS assessment once daily after their first flushing episode (if more than one happens to occur). The scale was from 0 to 3, where 0 represents no flushing, 1 represents mild flushing, 2 represents moderate flushing, and 3 represents severe flushing.
Time Frame: Up to Week 8
Population: PD Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants
  Baseline, No flushing | 17 | 14 | 9 | 18
  Week 2, No flushing | 15 | 17 | 18 | 19
  Week 4, No flushing | 12 | 17 | 15 | 20
  Week 6, No flushing | 14 | 14 | 14 | 20
  Baseline, Mild flushing | 1 | 1 | 6 | 0
  Week 2, Mild flushing | 1 | 1 | 1 | 0
  Week 4, Mild flushing | 1 | 0 | 1 | 0
  Week 6, Mild flushing | 0 | 0 | 1 | 0
  Baseline, Moderate flushing | 0 | 1 | 1 | 0
  Baseline, Severe flushing | 0 | 0 | 2 | 0

11. Secondary Outcome: Average Number of Flushing Episodes
Description: Flushing assessment was captured by participants in individual diaries provided to each study participant. Participants were instructed to return their diaries after each study visit (Week 2, Week 4, Week 6 and Week 8) where they were given a new diary for the time between visits. Participants with average number of flushing episodes was reported as "did not have flushing episode", "1 flushing episode", "2 flushing episode" and "3 or more flushing episode".
Time Frame: Up to Week 8
Population: PD Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants
  Did not have flushing episodes | 15 | 16 | 8 | 15
  1 flushing episode | 3 | 1 | 9 | 1
  2 flushing episode | 0 | 2 | 3 | 3
  3 or more flushing episode | 0 | 1 | 0 | 1

12. Secondary Outcome: Average Time to Onset of Flushing
Description: Flushing assessment was captured by participants in individual diaries provided to each study participant. Participants were instructed to return their diaries after each study visit (Week 2, Week 4, Week 6 and Week 8) where they were given a new diary for the time between visits. The time to the onset of the first flushing (if more than one happens to occur on each day) was analyzed.
Time Frame: Up to Week 8
Population: PD Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 12 | 5
Hours | 9.1 [6 to 13] | 3.6 [0 to 12] | 1.0 [0 to 9] | 4.1 [0 to 20]

13. Secondary Outcome: Participant's Average Duration of Flushing
Description: Flushing assessment was captured by participants in individual diaries provided to each study participant. Participants were instructed to return their diaries after each study visit (Week 2, Week 4, Week 6 and Week 8) where they were given a new diary for the time between visits. Participant's average duration of flushing was analyzed.
Time Frame: Up to Week 8
Population: PD Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 12 | 5
Minutes | 36.7 [5 to 90] | 151.7 [113 to 393] | 60.0 [4 to 160] | 72.1 [5 to 149]

14. Secondary Outcome: Number of Participants Who Withdrew Due to Flushing
Description: Flushing assessment was captured by participants in individual diaries provided to each study participant. Participants were instructed to return their diaries after each study visit (Week 2, Week 4, Week 6 and Week 8) where they were given a new diary for the time between visits.
Time Frame: Up to follow up (14 days from last dose)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Mean Episode of Flushing as Measured by Visual Analogue Scale (VAS)
Description: Flushing assessment was captured by participants in individual diaries provided to each study participant. Participants were instructed to return their diaries after each study visit (Week 2, Week 4, Week 6 and Week 8) where they were given a new diary for the time between visits. Participants self-assessed intensity of flushing using a 100 mm VAS once daily at the first flushing episode. The left hand side of the scale (0) represented 'No Flushing Sensation' and the right hand side of the scale (100) represented 'Unbearable Flushing Sensation'. The intensity of flushing of each episode was measured in centimeters (to the nearest 1/100) from the 0 point of the scale. Data is reported for average VAS scores over 8 weeks of treatment.
Time Frame: Up to Week 8
Population: PD Population was defined as all participants who provided PD data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 12 | 6
Scores on a scale | 9.0 (9.58) | 31.8 (19.24) | 24.9 (15.14) | 17.1 (26.76)

16. Secondary Outcome: Percent Change From Baseline in Fasting Plasma HDLc and Apolipoprotein A-I (ApoA1) Concentrations Over Eight Weeks of Administration With GSK256073 or Placebo
Description: Blood samples for analysis of fasting levels of HDLc and ApoA1 was collected at Baseline (Week 0) and Week 2, 4, 6 and 8. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the post-Baseline value from the Baseline value. Percent change from Baseline was calculated by multiplying change from baseline value with 100.
Time Frame: Baseline (Week 0) up to Week 8
Population: PD Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Percent change
  ApoA1, Week 2: number analyzed (Participants) | 18 | 19 | 19 | 20
  ApoA1, Week 2 | -2.7 (10.47) | -5.7 (15.45) | -5.9 (8.53) | -2.2 (8.63)
  ApoA1, Week 4: number analyzed (Participants) | 16 | 17 | 18 | 19
  ApoA1, Week 4 | 1.4 (8.73) | -1.8 (11.55) | -6.5 (11.01) | 1.3 (9.85)
  ApoA1, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 20
  ApoA1, Week 6 | 0.6 (14.23) | -3.1 (8.96) | -1.1 (9.75) | -1.3 (8.73)
  ApoA1, Week 8: number analyzed (Participants) | 16 | 15 | 15 | 19
  ApoA1, Week 8 | 4.2 (10.48) | -0.2 (13.50) | -2.0 (9.38) | 0.3 (9.25)
  HDLc, Week 2: number analyzed (Participants) | 18 | 19 | 19 | 20
  HDLc, Week 2 | -2.2 (10.50) | -8.4 (14.82) | -9.4 (13.76) | -2.8 (7.54)
  HDLc, Week 4: number analyzed (Participants) | 16 | 17 | 18 | 20
  HDLc, Week 4 | -1.2 (7.60) | -4.6 (19.54) | -7.0 (17.24) | -1.3 (8.00)
  HDLc, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 20
  HDLc, Week 6 | -2.0 (11.76) | -4.9 (12.80) | -7.9 (13.66) | 0.2 (11.17)
  HDLc, Week 8: number analyzed (Participants) | 16 | 15 | 15 | 20
  HDLc, Week 8 | 4.2 (12.99) | -1.9 (13.32) | -9.1 (15.46) | 1.1 (9.72)

17. Secondary Outcome: Percent Change From Baseline in Fasting Levels of Total Cholesterol (TC), Triglyceride (TG), Glucose, Low Density Lipoprotein Cholesterol (LDLc), Apolipoprotein A2 (ApoAII), Apolipoprotein B (ApoB) Over 8 Weeks of Administration With GSK256073 or Placebo
Description: Blood samples for analysis of fasting levels of TC, TG, glucose, LDLc, ApoAII and ApoB was collected at Baseline (Week 0) and Week 2, 4, 6 and 8. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the post-Baseline value from the Baseline value. Percent change from Baseline was calculated by multiplying change from baseline value with 100.
Time Frame: Baseline (Week 0) up to Week 8
Population: PD Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Percent change
  ApoAII, Week 2: number analyzed (Participants) | 14 | 17 | 18 | 19
  ApoAII, Week 2 | -9.9 (14.51) | -6.9 (13.60) | -4.7 (7.56) | 0.1 (17.22)
  ApoAII, Week 4: number analyzed (Participants) | 15 | 16 | 18 | 18
  ApoAII, Week 4 | 7.2 (38.06) | 3.4 (28.15) | -3.8 (11.36) | -1.6 (10.98)
  ApoAII, Week 6: number analyzed (Participants) | 15 | 15 | 16 | 19
  ApoAII, Week 6 | 5.9 (29.61) | -7.0 (10.96) | -5.3 (9.16) | 2.0 (15.60)
  ApoAII, Week 8: number analyzed (Participants) | 15 | 14 | 15 | 20
  ApoAII, Week 8 | 7.9 (30.30) | 5.2 (23.43) | 3.3 (27.68) | 2.1 (18.62)
  ApoB, Week 2: number analyzed (Participants) | 18 | 19 | 19 | 20
  ApoB, Week 2 | -8.1 (12.59) | -9.8 (9.42) | -2.2 (24.05) | -2.6 (7.58)
  ApoB, Week 4: number analyzed (Participants) | 16 | 17 | 18 | 19
  ApoB, Week 4 | -3.4 (8.85) | -6.1 (7.45) | 2.0 (22.30) | -0.8 (11.16)
  ApoB, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 20
  ApoB, Week 6 | -3.8 (11.51) | -6.5 (11.14) | 5.9 (26.74) | -1.8 (8.86)
  ApoB, Week 8: number analyzed (Participants) | 16 | 15 | 15 | 19
  ApoB, Week 8 | -2.8 (12.82) | -5.1 (12.14) | 6.5 (22.21) | -0.8 (8.37)
  Glucose, Week 2: number analyzed (Participants) | 18 | 19 | 19 | 20
  Glucose, Week 2 | 0.1 (8.74) | 7.0 (20.03) | 0.6 (13.64) | 2.8 (6.93)
  Glucose, Week 4: number analyzed (Participants) | 16 | 17 | 18 | 20
  Glucose, Week 4 | -0.3 (4.69) | 1.2 (10.50) | -2.2 (16.13) | 0.9 (8.68)
  Glucose, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 20
  Glucose, Week 6 | 0.7 (5.75) | 2.3 (13.37) | -2.6 (13.49) | 1.0 (9.79)
  Glucose, Week 8: number analyzed (Participants) | 16 | 15 | 15 | 20
  Glucose, Week 8 | -1.0 (10.19) | 2.6 (9.40) | -6.1 (14.98) | -0.0 (9.85)
  LDLc, Week 2: number analyzed (Participants) | 17 | 16 | 19 | 20
  LDLc, Week 2 | -2.7 (10.77) | -10.0 (12.24) | 2.1 (42.50) | -2.9 (12.08)
  LDLc, Week 4: number analyzed (Participants) | 16 | 15 | 18 | 19
  LDLc, Week 4 | -6.7 (6.19) | -7.4 (12.11) | 7.6 (50.51) | -3.0 (12.28)
  LDLc, Week 6: number analyzed (Participants) | 16 | 15 | 16 | 19
  LDLc, Week 6 | -4.3 (12.54) | -7.9 (11.85) | 7.7 (50.11) | 0.6 (13.09)
  LDLc, Week 8: number analyzed (Participants) | 16 | 13 | 15 | 19
  LDLc, Week 8 | -1.8 (12.25) | -6.5 (12.01) | 8.4 (50.73) | -3.0 (7.75)
  TC, Week 2: number analyzed (Participants) | 18 | 19 | 19 | 20
  TC, Week 2 | -4.0 (7.10) | -9.3 (8.28) | -3.3 (14.22) | -2.4 (6.58)
  TC, Week 4: number analyzed (Participants) | 16 | 17 | 18 | 20
  TC, Week 4 | -4.8 (5.28) | -5.9 (7.36) | -0.8 (12.57) | -2.5 (9.07)
  TC, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 20
  TC, Week 6 | -2.9 (8.63) | -6.2 (9.10) | -0.5 (13.54) | -1.3 (7.81)
  TC, Week 8: number analyzed (Participants) | 16 | 15 | 15 | 20
  TC, Week 8 | -0.5 (9.00) | -5.7 (8.96) | 1.3 (12.09) | -2.1 (5.49)
  TG, Week 2: number analyzed (Participants) | 18 | 19 | 19 | 20
  TG, Week 2 | 2.2 (32.06) | 16.9 (108.85) | 8.9 (48.90) | 6.6 (30.75)
  TG, Week 4: number analyzed (Participants) | 16 | 17 | 18 | 20
  TG, Week 4 | 6.1 (26.36) | 10.1 (55.36) | 3.0 (27.41) | 3.5 (24.63)
  TG, Week 6: number analyzed (Participants) | 16 | 16 | 16 | 20
  TG, Week 6 | 7.5 (21.81) | 0.9 (38.38) | 8.4 (23.84) | -4.6 (16.82)
  TG, Week 8: number analyzed (Participants) | 16 | 15 | 15 | 20
  TG, Week 8 | 6.6 (34.96) | 5.6 (41.75) | 21.0 (28.14) | -4.0 (17.76)

18. Secondary Outcome: Percent Change From Baseline in Insulin Over Eight Weeks of Administration With GSK256073 or Placebo
Description: Blood samples for analysis of insulin was collected at Baseline (Week 0) and Week 2, 4, 6 and 8. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the post-Baseline value from the Baseline value. Percent change from Baseline was calculated by multiplying change from Baseline value with 100.
Time Frame: Baseline (Week 0) up to Week 8
Population: PD Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Percent change
  Week 2: number analyzed (Participants) | 18 | 19 | 19 | 20
  Week 2 | 23.1 (82.20) | 21.2 (72.27) | 25.3 (92.41) | -2.8 (26.29)
  Week 4: number analyzed (Participants) | 16 | 17 | 18 | 20
  Week 4 | 9.1 (22.14) | 16.3 (73.97) | 13.2 (50.01) | -3.8 (22.33)
  Week 6: number analyzed (Participants) | 16 | 16 | 16 | 19
  Week 6 | 16.6 (43.40) | 17.8 (35.16) | 4.2 (44.83) | -3.4 (30.48)
  Week 8: number analyzed (Participants) | 16 | 15 | 15 | 20
  Week 8 | 2.8 (20.31) | 18.3 (47.56) | 13.7 (41.44) | -0.2 (29.89)

19. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) (Lp[a]) Over Eight Weeks of Administration With GSK256073 or Placebo
Description: Blood samples for analysis of Lp[a] was collected at Baseline (Week 0) and Week 2, 4, 6 and 8. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the post-Baseline value from the Baseline value. Percent change from Baseline was calculated by multiplying change from Baseline value with 100.
Time Frame: Baseline (Week 0) up to Week 8
Population: PD Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Percent change
  Week 2: number analyzed (Participants) | 11 | 10 | 14 | 12
  Week 2 | 1.8 (13.10) | -10.3 (13.52) | 4.5 (26.28) | -4.6 (14.91)
  Week 4: number analyzed (Participants) | 10 | 9 | 14 | 12
  Week 4 | -6.6 (20.62) | -11.3 (11.94) | 1.6 (19.33) | -1.7 (15.78)
  Week 6: number analyzed (Participants) | 11 | 10 | 12 | 12
  Week 6 | 2.7 (18.04) | -7.3 (16.50) | 6.5 (32.24) | -1.7 (13.73)
  Week 8: number analyzed (Participants) | 11 | 8 | 11 | 11
  Week 8 | 4.0 (13.56) | -15.8 (15.71) | 6.4 (18.87) | -5.6 (31.64)

20. Secondary Outcome: Percent Change From Baseline in Non-esterified Fatty Acids (NEFA) Over Eight Weeks of Administration With GSK256073 or Placebo
Description: Blood samples for analysis of NEFA was collected at Baseline (Week 0) and Week 2, 4, 6 and 8. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the post-Baseline value from the Baseline value. Percent change from Baseline was calculated by multiplying change from Baseline value with 100.
Time Frame: Baseline (Week 0) up to Week 8
Population: PD Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Percent change
  Week 2: number analyzed (Participants) | 18 | 19 | 19 | 20
  Week 2 | 32.1 (68.56) | 16.8 (53.84) | 29.1 (75.28) | 24.4 (44.56)
  Week 4: number analyzed (Participants) | 16 | 17 | 18 | 20
  Week 4 | 38.8 (70.88) | 37.4 (91.98) | 26.2 (80.52) | 7.0 (31.02)
  Week 6: number analyzed (Participants) | 16 | 16 | 16 | 19
  Week 6 | 47.8 (89.62) | 29.1 (73.47) | 8.0 (61.33) | -1.1 (28.66)
  Week 8: number analyzed (Participants) | 16 | 15 | 15 | 20
  Week 8 | 56.6 (112.49) | 59.4 (134.96) | 19.3 (60.35) | 10.4 (34.75)

21. Secondary Outcome: Plasma PK- Maximum Observed Concentration (Cmax)
Description: All participants treated with GSK256073 or placebo participated in PK sampling. Blood samples for PK analysis of GSK256073 to determine Cmax was collected at Week 2, 4, 6 and 8. For samples obtained during time windows, every attempt was made to collect three samples during each time window: pre-dose to 2 hours after dosing, 2 hours to 4.5 hours after dose, and 6 hours to 12 hours after dose. During each window, 3 samples spaced at least 30 minutes apart were collected (i.e., avoid collection from all participants at the same time within a window or only at the extremes of a time window). The first occurrence of the Cmax was determined directly from the raw concentration-time data.
Time Frame: 0-2 hours after dosing (pre-dose plus 3 samples spaced at least 30 minutes apart), 2 to 4.5 hours after dose (3 samples spaced at least 30 minutes apart) and 6-12 hours post dose (3 samples spaced at least 30 minutes apart) on Week 2, 4, 6 and 8
Population: PK Population was defined as all participants in the PK concentration population for whom PK parameters had been derived.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per mililiter (ng/mL)
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg
Number analyzed (Participants) | 15 | 15 | 17
Nanograms per mililiter (ng/mL) | 923.709 (128.18) | 7223.709 (35.09) | 22961.25 (62.36)

22. Secondary Outcome: Plasma PK- Time of Occurrence of Cmax (Tmax)
Description: All participants treated with GSK256073 or placebo participated in PK sampling. Blood samples for PK analysis of GSK256073 to determine Tmax was collected at Week 2, 4, 6 and 8. For samples obtained during time windows, every attempt was made to collect three samples during each time window: pre-dose to 2 hours after dosing, 2 hours to 4.5 hours after dose, and 6 hours to 12 hours after dose. During each window, 3 samples spaced at least 30 minutes apart were collected (i.e., avoid collection from all participants at the same time within a window or only at the extremes of a time window). The time at which Cmax was observed was determined directly from the raw concentration-time data.
Time Frame: as for outcome 21
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg
Number analyzed (Participants) | 15 | 15 | 17
Hours | 2.417 [0.50 to 7.73] | 1.350 [0.63 to 9.00] | 2.500 [0.50 to 25.98]

23. Secondary Outcome: Plasma PK- AUC(0-t)
Description: All participants treated with GSK256073 or placebo participated in PK sampling. Blood samples for PK analysis of GSK256073 to determine AUC(0-t) was collected at Week 2, 4, 6 and 8. For samples obtained during time windows, every attempt was made to collect three samples during each time window: pre-dose to 2 hours after dosing, 2 hours to 4.5 hours after dose, and 6 hours to 12 hours after dose. During each window, 3 samples spaced at least 30 minutes apart were collected (i.e., avoid collection from all participants at the same time within a window or only at the extremes of a time window). The AUC 0-t was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: as for outcome 21
Population: PK Analysis Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nanogram per milliliter (h*ng/mL)
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg
Number analyzed (Participants) | 15 | 15 | 16
Hour nanogram per milliliter (h*ng/mL) | 8352.281 (99.96) | 75587.96 (71.88) | 340551.4 (60.67)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected up to follow up (14 days from last dose).
Description: Safety population was used for the analysis of safety data.
Arm/Group | GSK256073 5 mg | GSK256073 50 mg | GSK256073 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 8/19 | 12/20 | 17/20 | 14/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK256073 5 mg (N=19) | GSK256073 50 mg (N=20) | GSK256073 150 mg (N=20) | Placebo (N=21)
Flushing (Vascular disorders) | 4 | 5 | 12 | 5
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 0/0 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Mean cell haemoglobin increased (Investigations) | 0 | 1 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Subgaleal haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was stopped for futility at the end of Part A due to lack of a compelling PK/PD relationship between GSK256073 and lipid effects that would predict success in achieving significant HDLc raising.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.